CLINICAL TRIAL: NCT06297356
Title: Investigation of the Effect of Stress Ball Utilisation on Treatment Duration, Dyspnoea Severity and Anxiety Level in Patients Receiving Nebuliser Therapy: A Randomised Controlled Study
Brief Title: The Effect of Stress Ball Utilisation on Treatment Duration, Dyspnea Severity and Anxiety Level in Nebuliser Therapy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kirsehir Ahi Evran Universitesi (Other)
Responsible Party: Principal Investigator, Yasemin CEYHAN, Assistant Proffesor, Kirsehir Ahi Evran Universitesi
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: YCEYHAN
Record Dates: First submitted 2024-02-20; First posted 2024-03-07 (Actual); Last update posted 2024-03-07 (Actual); Status verified 2024-02

CONDITIONS: Inhalation Therapy; Complications
Keywords: nebuliser; inhalers; dyspnea; anxiety level
MeSH Terms: conditions — Dyspnea

STUDY DESIGN:
Intervention Model Description: randomized controlled trial
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intervention (Experimental): This group will use a stress ball during nebuliser therapy. This process will be repeated at least twice a day.It will be a single application since the patients' current dyspnea and anxiety levels will be evaluated.
  Interventions: Device: Stress ball
- Control (No Intervention): Patients in this group will receive nebuliser therapy at least twice a day. However, no intervention will be made in the meantime. Measurements will be taken before and after any nebulizer treatment.

INTERVENTIONS:
Device: Stress ball — Stress balls are soft sponges with a diameter of 2-4 cm. The lightest starting level was preferred for the patients. Patients were allowed to take the stress ball in any hand they wanted. They were asked to squeeze and loosen the ball in their palm at 2-3 second intervals.
  Arms: intervention

SUMMARY:
Nebul Therapy is very effective in quickly improving the symptoms of respiratory system diseases. While applying this treatment, patients are expected to complete a sufficient period of time. However, this waiting and the symptoms of the disease may cause anxiety in the patient.

The aim of the study was to enable patients to spend their nebul period actively by using a stress ball. Thus, it was thought that it would make a positive contribution to dyspnea severity and anxiety levels.

The main questions it aims to answer are:

Does using a stress ball contribute positively to nebulizer usage time? Is the use of a stress ball effective in reducing the severity of dyspnea? Is using a stress ball effective in reducing anxiety levels?

For this purpose, participants will be asked to tighten and loosen the stress ball with one hand during the nebuliser therapy.

They will be expected to continue this with at least two nebuliser therapy per day. A control group will be used to determine the effectiveness of the stress ball. This group will not use a stress ball while receiving nebulizer treatment.

ELIGIBILITY:
Inclusion Criteria:

* Hospitalized for at least three days
* Having nebulizer treatment at least twice a day
* Medicines that have the same effect as prescribed (bronchodilators)
* Patients who are required to have at least 4 ml of medication in the reservoir
* Patients who have previous experience of using a nebulizer at home

Exclusion Criteria:

* Those who have severe exacerbation attacks
* People with speech problems
* People who experience severe dyspnea due to heart disease
* Those with high anxiety levels for any reason (death of a relative, etc.)
* Those with muscle or nerve problems in their hands
* Those who did not consent to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2023-10-01 (Actual); Primary Completion 2024-02-19 (Actual); Study Completion 2024-04-01 (Estimated)

PRIMARY OUTCOMES:
dyspnea severity | Through study completion, an average of 4 months.
  The patient's current dyspnea level is evaluated between 0-10. As it approaches 10, the intensity increases.
  The patient's dyspnea severity will be recorded before and after nebuliser therapy. This process will be done once.
anxiety levels | Through study completion, an average of 4 months.
  describes the patient's current anxiety level. The patient's current anxiety level is determined with the state anxiety scale developed for this purpose. The patient's anxiety levels will be recorded before and after nebuliser therapy. This process will be done once.
treatment duration | Through study completion, an average of 4 months.
  Defines the time between the start and end of nebuliser therapy. It is expected to be approximately 15-20 minutes. The patient's current condition will be measured. For this reason, it will be applied once.

SECONDARY OUTCOMES:
Vital signs: Respiratory rate | Through study completion, an average of 4 months.
  These are measurements that include the patient's respiratory rate. The patient's respiratory rate will be recorded before and after nebuliser therapy. This process will be done once.
Vital signs: Pulse | Through study completion, an average of 4 months.
  These are measurements that include the patient's pulse. The patient's vital signs will be recorded before and after nebuliser therapy. This process will be done once.
Vital signs: Blood pressure | Through study completion, an average of 4 months.
  These are measurements that include the patient's blood pressure. The patient's vital signs will be recorded before and after nebuliser therapy. This process will be done once.
saturation | Through study completion, an average of 4 months.
  It is the percentage of oxygen saturation of the blood. Measured with a probe from the finger. The patient's saturation levels will be recorded before and after nebuliser therapy. This process will be done once.

CONTACTS AND LOCATIONS:
Locations (1):
- Yasemin CEYHAN, Kırşehir, Center, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No